CLINICAL TRIAL: NCT03047811
Title: The Study of Targeted NY-ESO-1 T Cell Receptor (TCR) Genetic Modified Autologous T Cells Treatment of Advanced Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xianghua Wu, Clinical Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NY-TCR WXH 2016
Record Dates: First submitted 2017-01-25; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Advanced Malignant Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR - T cell therapy (Experimental): Peripheral blood mononuclear cells collected: draw 100-150 ml of peripheral blood in patients and separate of the peripheral blood mononuclear cells, the total number of cells 1.5 * 10 ^ 7 / kg - 1 * 10 ^ 8 / kg Fludarabine 25 mg/m2 + NS 250 ml, ivgtt qdx5d, CTX 60 mg/kg + NS 250 ml, ivgtt qd x2d, should be in front of the TCR - T cells infusion of 4 days reinfusion the total number of T cells （1* 10 ^ 8 / kg - 10 * 10 ^ 8 / kg） in 3 days , infusion 10-15 minutes, should not be more than 20 minutes.
  Interventions: Other: TCR - T cell therapy

INTERVENTIONS:
Other: TCR - T cell therapy — Low dose group: 1 x 10 ^8 /kg T cell total reinfusion. High dose groups: 10 x 10 ^ 8 / kgT cell total reinfusion.

SUMMARY:
The study of targeted NY-ESO-1 T cell receptor (TCR) genetic modified autologous T cells treatment of advanced solid tumors

1. The main purpose - security and ORR;
2. A secondary purpose - median progression-free surial;1 year, 2 years, total 5 years survival rate;The quality of life.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 volunteered for the clinical research and signed informed consent. 3.1.2 aged 18-70, expected lifetime > 3 months. 3.1.3 gender not limited. 3.1.4 late lung cancer (stage IIIb/IV), (IV) with esophageal carcinoma, and melanoma (advanced), no other effective cure Treatment method can be selected patients. 3.1.5 biopsy IHC confirmed positive expression, NY - ESO - 1 or 50% of the tumor cells IHC staining in 2 + and/or 3 +.Organization based on time in the group in the year before, can be a tumor tissue, can also be a pleural effusion cells

Exclusion Criteria:

3.2.1 this study used in the process of cell preparation ingredients allergy, such as penicillin, streptomycin.

3.2.2 used within a week of tyrosine kinase inhibitors (the treatment such as, for it), or other cancer drugs.

3.2.3 is systemic anti-cancer therapy, including immune therapy, such as accept the immune cells within a month back to lose Therapy or biological treatment.6 weeks used cancer associated with tumor immune single resistance (including the PD, PD - L1 and - 1 CTLA 4 single resistance). 3.2.4 have vital organs, such as cardiovascular, respiratory system disease, myocardial infarction, myocardial ischemia, the coronary artery bypass History or coronary ischemia symptoms, obstructive or restrictive lung disease. 3.2.5 the patient's immune tolerance is poor, may on the immune cells in treatment of the reaction of low or prone to toxic reactions.

3.2.6 always have autoimmune and immunodeficiency disease. 3.2.7 radiation pneumonitis. 3.2.8 depends on oxygen. 3.2.9 four weeks into the set of other therapeutic studies or clinical trials. 3.2.10 used experimental vaccine in two months 3.2.11 systemic corticosteroids used within two weeks, hydroxyurea or immune inhibitors (such as IL - 2, Interferons alpha, IFN - gamma, GSF, mTOR inhibitors, ring spore element, etc.).Recently or are using suction The sex hormone. 3.2.12 year have chronic or recurrent severe autoimmune diseases. 3.2.13 uncontrolled active infection. 3.2.14 2-4 acute or persistent during graft versus host disease (GVHD). 3.2.15 serious heart disease, after treatment of the disease is still unstable, into the group of the first six months after myocardial infarction, and congestion Heart failure, unstable angina, symptoms of pericardial effusion or unstable arrhythmia.

3.2.18 always suffer from other cancers, but does not include: A. basal cell carcinoma and squamous cell carcinoma after active treatment, the wound healed completely.

B. the cervical or breast carcinoma in situ cure for at least three years. C. primary malignant tumors were removed completely, completely relieve five years or more.

3.2.19 accompanied by primary or secondary brain tumor patients. 3.2.20 the mentally disabled. 3.2.21 doubt or have alcohol and drug abuse history. 3.2.22 physicians determine cannot or may not be able to complete the test subjects.

3.2.23 any not listed may interfere with the patient to participate in the active disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-08-26 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | From date of randomization until the date of date of death from any cause, whichever came first, assessed up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No